CLINICAL TRIAL: NCT03653819
Title: High Intensity Interval Training (HIIT) on Stationary Bike With and Without Compression Stockings for Patients With Cancer-related Lymphedema in the Lower Limbs - a Feasibility Study
Brief Title: High Intensity Interval Training (HIIT) for Patients With Cancer-related Lymphedema in the Lower Limbs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Merete Celano Wittenkamp, Pricipal Investigator, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Lympha feasibility
Record Dates: First submitted 2018-08-23; First posted 2018-08-31 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Lymphedema of Leg; Cancer of Cervix; Cancer, Ovarian; Cancer, Endometrial; Cancer of the Prostate; Malignant Melanoma
Keywords: Compression Stockings; Feasibility Study; Physical Activity; High Intensity Interval Training; Cross over trial
MeSH Terms: conditions — Uterine Cervical Neoplasms; Ovarian Neoplasms; Endometrial Neoplasms; Prostatic Neoplasms; Melanoma; Motor Activity

STUDY DESIGN:
Intervention Model Description: All participants complete a baseline assessment followed by the randomisation to HIIT + compression or HIIT - compression.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT + compression (Other): 2 sessions of High Intensity Interval Training (HIIT) on a stationary bike. First exercise session with compression garments/second without.
  Interventions: Other: First exercise session + compression
- HIIT - compression (Other): 2 sessions of High Intensity Interval Training (HIIT) on a stationary bike. First exercise session without compression garments/second with
  Interventions: Other: First exercise session - compression

INTERVENTIONS:
Other: First exercise session + compression — The Interval Training consists of a 5 minute warm-up on the stationary bike followed by 7 intervals of cycling for 1 minute at level 15-16 on the Borg Scale of Perceived Exertion. Inbetween intervals, participants reduce resistance on the stationary bike and pedals for 1 minute at level 11-12 on the Borg Scale. The session ends with a 5-10 minute cool-down pedaling and stretching exercises for the lower limbs.
  Arms: HIIT + compression
Other: First exercise session - compression — The Interval Training consists of a 5 minute warm-up on the stationary bike followed by 7 intervals of cycling for 1 minute at level 15-16 on the Borg Scale of Perceived Exertion. Inbetween intervals, participants reduce resistance on the stationary bike and pedals for 1 minute at level 11-12 on the Borg Scale. The session ends with a 5-10 minute cool-down pedaling and stretching exercises for the lower limbs.
  Arms: HIIT - compression

SUMMARY:
The aim of the study is to explore the feasibility and safety of High Intensity Interval Training on a stationary bike for patients with lymphedema in the lower limbs and the role of compression garments during exercise.

The design of the study is a cross-over randomized clinical trial. Participants will be randomized into two groups. Both will perform two separate exercise sessions.Group A will perform the first exercise with compression garment and the second session without compression garment, with wash-out period of 1 week between sessions. Group B will perform the exercise sessions in the opposite order.

DETAILED DESCRIPTION:
Lymphedema is a condition afflicting cancer patients who undergo surgery with removal of lymph nodes, chemotherapy and radiation. Lymphedema is a consequence of impaired lymphatic drainage in the interstitium, which causes edema and inflammation in the subcutaneous tissue. The symptoms are swelling, puffiness, tightness, heaviness and pain in the affected area.

Lymphedema can be reduced by complete decongestive therapy, which consists of skin care, manual lymphatic drainage, compression bandaging and exercise. At the end of treatment, patients are provided with custommade compression garments to be worn during daytime in order to maintain the reduction in the edema.

Lymphedema has a negative impact on activities of daily living and health-related quality of life. Patients with lymphedema should be encouraged to engage in physical activity despite their condition in order to prevent relapse of cancer and development of other diseases. Likewise physical activity helps to maintain a healthy weight, which is important as obesity has a negative impact on lymphedema. The lymphatic system is also stimulated by physical activity and exercise and can reduce the symptoms from the lymphedema.

Several studies have been published on the safety and benefits of exercise for women with breastcancer related lymphedema. However, only a few studies have investigated the feasibility of exercise to patients with lymphedema in the lower limbs. Also the role of compression garments during exercise have not been throughly explored.

ELIGIBILITY:
Inclusion Criteria:

* unilateral or bilateral lymphedema in the lower limbs
* secondary lymphedema
* wears custommade compression stockings during daytime
* lymphedema in stage 1, 2A or 2B (Classification from the International Society of Lymphology)
* legally competent persons with ability to read and understand Danish.

Exclusion Criteria:

* inability to perform the intervention, as assessed by the person performing inclusion.
* lymphedema in stage 0 or 3 (Classification from the International Society of Lymphology)
* ongoing complete decongestive lymphedema therapy
* untreated erysipelas
* ongoing oncologic treatment: chemotherapy, radiation, immune therapy,
* known metastatic cancer
* comorbidities e.g. deep venenous thrombosis, serious heart disease, renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2018-11-13 (Actual)

PRIMARY OUTCOMES:
Feasibility rate | After 3 months
  Number of invited eligible participants enrolled in the study
Completion rate | After 3 months
  Number of enrolled participants completing both interventions

SECONDARY OUTCOMES:
Participant satisfaction | Week 2
  At the end of the study participation, data describing participant satisfaction will be collected to answers questions on acceptability. All participants will be given a questionnaire and will be asked to rank various aspects of the intervention including exercising without compression garments "as not at all satisfied", "not very satisfied", "somewhat satisfied" or "very satisfied". Feasibility will be defined as >75% of participants reporting they are "very" or "somewhat satisfied" with the intervention.
Change in pain related to lymphedema | Hour 0 and 1 post each exercise sessions
  Participant-reported pain measured on a numeric range scale 0-10, "0" indicating no pain and "10" as worst imaginable pain. Measurements will be made immediately before and after each exercise session.
Change in tension related to lymphedema | Hour 0 and 1 post each exercise sessions
  Participant-reported tension measured on a numeric range scale 0-10, "0" indicating no tension and "10" worst imaginable tension. Measurements will be made immediately before and after each exercise session.
Change in heaviness related to lymphedema | Hour 0 and 1 post each exercise sessions
  Participant-reported heaviness measured on a numeric range scale 0-10, "0" indicating no heaviness and "10" worst imaginable heaviness. Measurements will be made immediately before and after each exercise session.
Change in volume of lower limbs | Hour 0 and hour 1 post each exercise sessions
  Tape Measurements(cm) at 8 cm intervals, converted to volume (ml) by formula of truncated cone. Measurements will be made immediately before and after each exercise session
Change in extracellular fluid in the lower limbs | Hour 0 and hour 1 post each exercise session
  Bioimpedance Spectroscopy. Measurements will be made immediately before and after each exercise session.
Change in weight of the lower limbs | Hour 0 and hour 1 post each exercise session
  Dual Energy Xray Absorptiometry, a full body scan is performed. Afterwards regions of interest is marked and weight of each lower limb calculated. Measurements will be made immediately before and after each exercise session.

CONTACTS AND LOCATIONS:
Overall Officials: Merete C Wittenkamp, PT, Principal Investigator — Department of Physiotherapy and Occupational Therapy at Herlev and Gentofte Hospital,; Carsten B Juhl, PT MPH PhD, Study Chair — Department of Physiotherapy and Occupational Therapy, Herlev and Gentofte Hospital/Research Unit for Musculoskeletal Function and Physiotherapy, University of Southern Denmark.; Anders Vinther, PT MSc PhD, Study Chair — Department of Physiotherapy and Occupational Therapy, Herlev and Gentofte Hospital
Locations (1):
- Department of Physiotherapy and Occupational Therapy, Herlev and Gentofte Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wittenkamp MC, Juhl CB, Zerahn B, Vinther A. Exercise and cancer-related lymphedema in the lower limbs-a randomized cross-over trial on high-intensity interval training (HIIT) with and without compression garments. Support Care Cancer. 2025 Apr 16;33(5):391. doi: 10.1007/s00520-025-09458-x. PMID 40240614